CLINICAL TRIAL: NCT02064322
Title: SAIF: Sacroiliac Fusion Study Using the Zyga SImmetry Sacroiliac Joint Fusion System
Brief Title: SAIF: Sacroiliac Fusion Study
Acronym: SAIF
Status: Terminated | Type: Observational
Sponsor: Zyga Technology, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLP 007-001
Record Dates: First submitted 2014-02-12; First posted 2014-02-17 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Sacroiliac Joint Dysfunction
Keywords: sacroiliac joint fusion; SIJ fusion; SI joint

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SImmetry Implant: Subjects who are indicated for the SImmetry Device according to the approved product labeling and inclusion/exclusion criteria will receive a SImmetry implant.
  Interventions: Device: SImmetry Implant

INTERVENTIONS:
Device: SImmetry Implant — The SImmetry system is commercially available. The implanted devices consist of a range of thread-tapping cannulated implants designed to transfix the sacrum and ilim, providing stability for intra-articular fusion.
  The SImmetry Surgical Instruments include standard manual surgical instruments used to access and prepare the sacroiliac joint space for intra-articular fusion.

SUMMARY:
The purpose of the SAIF study is to evaluate the SImmetry Sacroiliac Joint Fusion System for fusion and pain reduction of the SI joint.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, single center study to collect data on fusion and pain reduction following implantation of the SImmetry device. Up to 15 total subjects will be implanted and followed for 24 months. Data will be collected pre-operatively, at implant, discharge, and at specified follow-up time points (6 weeks, 3 months, 6 months, 12 months, 24 months.)

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be indicated for the SImmetry device according to the approved SImmetry labeling
* Subject has three (3) positive (experiences pain) Provocative Tests for SIJ pain; for example, Compression, Thigh Thrust, FABER, Distraction or Gaenslen's
* Subject has documentation of failed, non-operative management of SIJ pain for ≥ 6 months prior to surgery; for example, use of medications, braces, SI belts, orthotics, physical therapy or manual manipulation
* The subject has one (1) positive diagnostic SIJ injection, resulting in a ≥50% decrease in pain from the anesthetic portion of the injection
* The subject has VAS back pain score of ≥ 60 mm
* The subject has an ODI ≥ 40%
* The subject is at least 18 years of age and skeletally mature
* The subject agrees and is able to comply with study requirements

Exclusion Criteria:

* Subjects contraindicated per the cleared labeling will be excluded from participation in the study
* The subject has pelvic soft tissue or bony tumors
* The subject has had any trauma causing fracture of the sacrum or iliac bones or has had spinal trauma leading to a neurological deficit
* The subject has a history of a central nervous system (CNS) disorder(s)
* The subject is pregnant or is planning on becoming pregnant in the next two years
* The subject has chemical dependency problems as evidenced by a history of drug abuse which is documented in their past medical history or is elicited from an interview
* The subject has a history of significant emotional or psychosocial disturbance (anxiety attacks, obsessive/compulsive disorders, depression or schizophrenia) as documented in their past medical history or elicited by an interview

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the Investigator's standard patient population diagnosed with SIJ pain and representing candidates' for SIJ fusion.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2014-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
SI Joint Fusion | 12 months
  Confirmed fusion of the SI joint at 12 and 24 months, defined as as presence of a continuous segment of solid bridging bone that extends from the sacrum to the ilium.
SI Joint Pain Reduction | 6 months
  SI joint pain reduction evaluated by use of Visual Analogue Scale (VAS) for back pain for comparison of baseline to 6 months.

SECONDARY OUTCOMES:
SI Joint Pain Reduction | 12 and 24 months
  SI joint pain reduction evaluated by use of Visual Analogue Scale (VAS) for back pain for comparison of baseline to all follow-up visits.